CLINICAL TRIAL: NCT01364532
Title: A Randomized Study of Transradial Versus Transulnar Artery Approach for Coronary Interventions
Brief Title: Transradial Versus Transulnar Artery Approach for Coronary Interventions
Acronym: AURA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Patras (Other)
Responsible Party: George Hahalis, Patras University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-5
Record Dates: First submitted 2011-05-27; First posted 2011-06-02 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-04

CONDITIONS: Arterial Access in Percutaneous Coronary Angiography or Intervention
Keywords: transulnar arterial access; transradial arterial access; percutaneous coronary intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transulnar arterial access (Experimental): Transulnar arterial access for coronary angiography, ad-hoc or elective PCI
  Interventions: Procedure: Transulnar arterial access
- Transradial arterial access (Active Comparator): Transradial arterial access for coronary angiography, ad-hoc or elective PCI
  Interventions: Procedure: Transradial arterial access

INTERVENTIONS:
Procedure: Transulnar arterial access — Transulnar arterial access in coronary angiography, ad-hoc or elective PCI
  Arms: Transulnar arterial access
Procedure: Transradial arterial access — Transradial arterial access for coronary angiography,ad-hoc or elective PCI
  Arms: Transradial arterial access

SUMMARY:
The transradial route is increasingly used as an access site in percutaneous coronary interventions, as it is considered equivalent to transfemoral approach in terms of efficacy but with a decreased vascular complication risk. Information concerning the efficacy and safety of transulnar approach is sparse. This is a prospective, randomized, investigator-initiated study to compare transradial versus transulnar approach as a default strategy for coronary angiography, ad-hoc or elective percutaneous coronary intervention (PCI). Consecutive eligible patients with an indication for coronary angiography, will be randomized after written informed consent in a 1:1 ratio to either transradial or transulnar access. Assessment of angiographic and procedural characteristics(including amount of contrast medium, arterial access, fluoroscopy and procedural time), as well as any vascular or other peri-procedural complications of the cases enrolled, will be performed. After hospital discharge, all patients will return at Day 60 ±5 days for Doppler ultrasound assessment of the forearm vessels and documentation of major adverse cardiovascular events (defined as death, myocardial infarction, target vessel revascularization and stroke. Coronary angiography patients will be additionally randomized in a 1:1 ratio to either 2500 or 5000 IU of unfractioned heparin.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Plan for Coro- and ad hoc PCI, if necessary
* Written informed consent

Exclusion Criteria:

* Cardiogenic shock, haemodynamic instability, Killip class III
* Chronic hemodialysis
* Coronary artery bypass grafting (CABG) with either bilateral internal mammary artery (IMA) or bilateral radial artery use

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Successful arterial access free from need for crossover and free from vascular or coronary ischemic complications (MACEs)within 60± days | The primary end point will be assessed within 60±5 days after randomization
  MACEs are considered both vascular and coronary ischemic complications. Vascular complications include arterial occlusion, local arterial perforation, compartment syndrome, pseudoaneurysm, fistula formation, major bleeding, hematoma of at least 10cm length, or any vascular damage requiring prolonged hospitalization or intervention.
  Coronary ishcemic complications include cardiac death, non fatal myocardial infarction, urgent repeat revascularization and stroke.

SECONDARY OUTCOMES:
Fluoroscopy time | Fluoroscopy time will be assessed within 1 minute after the end of coronary angiography or coronary intervention
  Fluoroscopy time (in seconds) assessed within 1 minute after the end of coronary angiography or coronary intervention
Amount of contrast medium | The amount of contrast medium will be assessed within 1 minute after the end of coronary angiography or coronary intervention
  Volume of contrast medium (ml) will be assessed within 1 minute after the end of coronary angiography or coronary intervention
Vascular complication defined as post-procedural occlusion, perforation, pseudo-aneurysm, fistula or hematoma formation | Vascular complication will be assessed 6 hours after the end of coronary angiography or intervention
  Vascular complication (defined as post-procedural occlusion, perforation, pseudo-aneurysm, fistula or hematoma formation of at least 10 cm length, compartment syndrome) will be assessed 6 hours after the end of coronary angiography or intervention
Procedural duration (defined as the sum of arterial access, coronary angiography and coronary intervention duration) | Procedural duration will be assessed within 1 minute after the end of coronary angiography or coronary intervention
  Procedural duration (defined as the sum of arterial access, coronary angiography and coronary intervention duration)will be assessed within 1 minute after the end of coronary angiography or coronary intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Patras University Hospital, Pátrai, Rion, Greece

REFERENCES:
- [Derived] Hahalis G, Tsigkas G, Xanthopoulou I, Deftereos S, Ziakas A, Raisakis K, Pappas C, Sourgounis A, Grapsas N, Davlouros P, Galati A, Plakomyti TE, Mylona P, Styliadis I, Pyrgakis V, Alexopoulos D. Transulnar compared with transradial artery approach as a default strategy for coronary procedures: a randomized trial. The Transulnar or Transradial Instead of Coronary Transfemoral Angiographies Study (the AURA of ARTEMIS Study). Circ Cardiovasc Interv. 2013 Jun;6(3):252-61. doi: 10.1161/CIRCINTERVENTIONS.112.000150. Epub 2013 Jun 4. PMID 23735472